CLINICAL TRIAL: NCT00599092
Title: Pituitary Tumor Surveillance: Pathogenetic Correlation
Brief Title: Pituitary Tumor Surveillance: Pathogenic Correlation
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Shlomo Melmed, MD, Professor of Medicine, Cedars-Sinai Medical Center
Other Study IDs: 2873; 2873
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pituitary Tumor
Keywords: pituitary tumor; recurrence
MeSH Terms: conditions — Pituitary Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to observe predictors of pituitary tumor recurrence and markers of persistent disease activity in patients harboring pituitary mass lesions of all types.

DETAILED DESCRIPTION:
The purpose of this study is to observe predictors of pituitary tumor recurrence and markers of persistent disease activity through computerized collection of comprehensive demographic, therapeutic, pathologic and outcome information on patients harboring pituitary mass lesions of all types.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed pituitary disease

Exclusion Criteria:

* patients who do not have confirmed pituitary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 1997-01; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center, Pituitary Center
Locations (1):
- Cedars-Sinai Medical Center, Pituitary Center, Los Angeles, California, United States